CLINICAL TRIAL: NCT05132764
Title: Effect of Micro-osteo-perforations on the Rate of Alignment of Mandibular Anterior Teeth.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Shahida Jehan, Dr, Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC : 2021-06-070
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Orthodontics
Keywords: Microosteoperforations; Little's index; Rate of tooth movement

STUDY DESIGN:
Intervention Model Description: Two parallel arm randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor and the investigator will have no knowledge of the intervention in the digital models.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOPs group (Experimental): Orthodontic treatment will be started in all subjects using fixed preadusted edgewise appliance (0.022-in MBT prescription, Ortho Organizers, Inc. USA).Local anesthesia will be given in lower arch .Two points for screw insertion will be demarcated on buccal mucosa, in each interdental segment using a calibrated periodontal probe. Orthodontic miniscrew (AbsoAnchor, Korea) of 1.3 mm diameter will be used for MOPs to the depth of 2-3 mm into the buccal cortical bone. An endodontic rubber stopper will be set for required / optimal depth on miniscrew and MOPs will be performed. After the intervention, the patients will be instructed for maintaining good oral hygiene and to take analgesics, such as acetaminophen, only if necessary.
  Interventions: Procedure: Microosteoperforations
- Control group (No Intervention): Orthodontic treatment will be started in all subjects using fixed preadusted edgewise appliance (0.022-in MBT prescription, Ortho Organizers, Inc. USA).The control group will receive no MOPs at the alignment stage.

INTERVENTIONS:
Procedure: Microosteoperforations — 2 inter radicular bone microosteoperforations using temporary anchorage device tip.
  Arms: MOPs group

SUMMARY:
Micro osteoperforation is an easy, safe and effective method of accelerating orthodontic tooth movement by 2-3 times.it has been reported to increased the osteoblastic activity and some acceleration of the rate of canine retraction,reducing the treatment duration and associated side effects. The aim of this study is to assess the effect of MOPs on the rate of alignment of mandibular anterior teeth.

DETAILED DESCRIPTION:
MATERIAL AND METHODS:

STUDY DESIGN: Two parallel arm randomized controlled clinical trial SETTING: Orthodontics Department, Rehman College of Dentistry. DURATION OF STUDY: one year SAMPLING TECHNIQUE: non-probability consecutive sampling.

SAMPLE SELECTION:

INCLUSION CRITERIA

1. Malocclusion cases with mandibular anterior segment crowding.
2. Age range 13-30 years.

EXCLUSION CRITERIA:

1. Missing lower anterior tooth.
2. Systemic diseases/Medications affecting bone biology.
3. Previous orthodontic treatment.
4. Poor oral hygiene status.
5. Active periodontal disease
6. Syndromes. DATA COLLECTION Written informed consent from the patients will be taken after clarification of the purpose of the intervention and the associated risks and benefits. Orthodontic treatment will be started in all subjects using fixed preadusted edgewise appliance (0.022-in MBT prescription, Ortho Organizers, Inc. USA). After bonding of lower arch the patients will be randomized into control and experimental groups.

Patients will be randomly allocated, through computer generated tables in Microsoft Excel Software, into parallel groups with a 1:1 allocation ratio. Allocation will be concealed in opaque envelopes and opened only at the time of intervention.

Local anesthesia will be given in lower arch on each side approximately 1cm from labial frenum. Two points for screw insertion will be demarcated on buccal mucosa, in each interdental segment, by bleeding points using a calibrated periodontal probe. Probe tip will be inserted to the level of bone to measure the thickness of gingiva. The measurement will be added to the depth of perforation needed i-e 2 - 3 mm into the bone. First point will be marked at a distance of 3mm from free gingival margin and second point will be marked 3mm from the first one. Orthodontic miniscrew (AbsoAnchor, Korea) of 1.3 mm diameter will be used for MOPs to the depth of 2-3 mm into the buccal cortical bone. An endodontic rubber stopper will be set for required / optimal depth on miniscrew and MOPs will be performed. After the intervention, the patients will be instructed for maintaining good oral hygiene and to take analgesics, such as acetaminophen, only if necessary.

The control group will receive no MOPs at the alignment stage. Alignment will be started in both control and experimental groups using 0.012 NiTi (North American Braces, USA). Both the groups will be followed every month for maximum six months. Digital scan of lower arch will be taken on each visit. Each scan will be labelled for identification, date of scan taking and little index score .For reliability 20 randomly selected scan will be rescored for little index by the same examiner as well as another examiner after 2 weeks for intra and inter-examiner reliability.

ELIGIBILITY:
Inclusion Criteria:

1. Malocclusion cases with mandibular anterior segment crowding.
2. Age range 13-30 years.

Exclusion Criteria:

1. Missing lower anterior tooth.
2. Systemic diseases/Medications affecting bone biology.
3. Previous orthodontic treatment.
4. Poor oral hygiene status.
5. Active periodontal disease
6. Syndromes

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of alignment of lower anterior teeth | 6 months
  Rate of alignment of lower anterior teeth

SECONDARY OUTCOMES:
clinical crown length | 6 moths
  clinical crown length

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad K Asif, PhD, Study Director — Rehman Medical Institute
Locations (1):
- Sohrab Shaheed, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No